CLINICAL TRIAL: NCT02364310
Title: Evaluation médico-économique de la Stimulation unilatérale du Sinus Carotidien Dans le Traitement de l'Hypertension artérielle résistante: Essai Multicentrique contrôlé, randomisé, Ouvert Avec évaluation d'efficacité Tensionnelle et de sécurité
Brief Title: Economic Evaluation of Baroreceptor STIMulation for the Treatment of Resistant HyperTensioN
Acronym: ESTIM-rHTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pr Patrick ROSSIGNOL (Other)
Responsible Party: Sponsor-Investigator, Pr Patrick ROSSIGNOL, PU-PH, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00632-45
Record Dates: First submitted 2015-02-02; First posted 2015-02-18 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Hypertension
Keywords: Hypertension; baroreceptor stimulation; Hypertension resistant
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baroreceptor stimulation on top of the best medical care (Experimental): Baroreceptor stimulation with Barostim Neo TM
  Interventions: Device: Baroreceptor stimulation with Barostim Neo TM
- Best medical care (No Intervention): Best medical care

INTERVENTIONS:
Device: Baroreceptor stimulation with Barostim Neo TM
  Arms: Baroreceptor stimulation on top of the best medical care

SUMMARY:
Medico-economics assessment (cost-effectiveness) of the unilateral carotid barostimulation with Barostim NeoTM compared to usual care in patients with resistant hypertension (multicenter randomized, PROBE trial), followed-up for 12 months, with a lifetime-long modeling.

ELIGIBILITY:
Main inclusion Criteria:

* 18-85 years old men or women
* Resistant hypertension on 4 medications incl. thiazide or thiazide-like diuretics at appropriate doses + spironolactone (unless spironolactone intolerance)
* Essential hypertension documented (bilan < 2 years old)
* eGFR ≥ 30 ml/min/1,73 m2
* No carotid condition associated with a contra-indication for Barostim NeoTM use

Main exclusion Criteria:

* Patients with documented secondary hypertension, besides Obstructive Sleep Apnea
* Symptomatic orthostatic hypotension
* Patient with prior syncope or myocardial infarction, unstable angina pectoris, or cerebrovascular within 3 months before inclusion
* Patient with type 1 diabetes mellitus
* Patient with permanent atrial fibrillation
* Patient with brachial circumference of ≥ 46cm
* Patient with BMI>45kg/m2
* Pregnancy, breastfeeding or planning a pregnancy within 2 years
* NeoTM implantation anatomic contra-indications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
12th month diurnal SBP (mmHg) measured on ABPM, adjusted on baseline SBP, also used to compute the incremental cost-effective ratio (to identify the extra cost of unilateral carotid barostimulation in BP reduction compared to usual care) | 12 months

SECONDARY OUTCOMES:
Mean SBP 24h on ABPM (mmHg) | 6 and 12 months
  Comparison with usual care
Mean nocturnal SBP on ABPM (mmHg) | 6 and 12 months
  Comparison with usual care
Mean DBP 24h on ABPM (mmHg) | 6 and 12 months
  Comparison with usual care
Mean diurnal DBP on ABPM (mmHg) | 6 and 12 months
  Comparison with usual care
Mean nocturnal DBP on ABPM (mmHg) | 6 and 12 months
  Comparison with usual care
Casual SBP (mmHg) | 6 and 12 months
  Comparison with usual care
Casual DBP (mmHg) | 6 and 12 months
  Comparison with usual care
Casual PP (mmHg) | 6 and 12 months
  Comparison with usual care
Pulse wave velocity (m/s) | 6 and 12 months
  Comparison with usual care
Central Pulse Pressure (mmHg) | 6 and 12 months
  Comparison with usual care
Function and Left ventricular mass on echocardiography (g/m²) | 6 and 12 months
  Comparison with usual care
Evolution of the kidney function (eGFR - MDRD - ml/min/1.73 m²) | 6 and 12 months
  Comparison with usual care
Microalbuminuria (mg/mmol creatinine) | 6 and 12 months
  Comparison with usual care
Antihypertensive regimen (Number of antihypertensive drugs) | 6 and 12 months
  Comparison with usual care
EuroQol5D (score) | 6 and 12 months
  Comparison with usual care
Cardiovascular events (number of events) | baseline, 6 and 12 months
  Comparison with usual care
Global cardiovascular risk (scale) | 6 and 12 months
  Comparison with usual care
Surgery Morbidity | 1 month
  Clavien Dindo Scale, morbidity 1 month after surgery
cerebrovascular events (number of events) | baseline, 6 and 12 months
  Comparison with usual care
kidney events (number of events) | baseline, 6 and 12 months
  Comparison with usual care

OTHER OUTCOMES:
Cost of unilateral carotid barostimulation including hospital stay | participants will be followed for the duration of hospital stay, an expected average of 2 days
ICER: difference in cost / difference in office systolic blood pressure (SBP) in mmHg | 12 months
ICER/ICER: difference in cost / difference in QALY (quality-of-life-adjusted survival based on the clinical trial data and the modeling results) for the lifetime modeling | 12 months
Budget impact (cost in Euros) | 4 years
Number of outpatient visits for hypertension management in both groups | 12 months
Morbidity | 6 and 12 months
  Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Patrick ROSSIGNOL, Prof, Principal Investigator — CHRU Nancy; Michel AZIZI, Prof, Principal Investigator — APHP-HEGP
Locations (15):
- France (15):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Arthur Gardiner, Dinard
  - CHU de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Hospices civils de Lyon, Lyon
  - APHM, Marseille
  - CHRU de Nancy, Nancy
  - APHP -Hotel Dieu hospital, Paris
  - GH la Pitié Salpêtrière, Paris
  - HEGP, Paris
  - CHU de Poitiers, Poitiers
  - CHU de RENNES, Rennes
  - CHU de Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
  - CHRU de Tours, Tours